CLINICAL TRIAL: NCT01786876
Title: A Phase 1 Study to Investigate the Absorption, Metabolism and Excretion of [14C]SPD557 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Adsorption, Metabolism and Excretion (AME) of Single Dose Radiolabeled SPD557 in Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SPD557-107
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
Keywords: Radiolabelled; AME

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiolabeled SPD557 (Experimental)
  Interventions: Drug: Radiolabeled SPD557

INTERVENTIONS:
Drug: Radiolabeled SPD557 — A single oral dose of 2 mg radiolabeled SPD557 administered on Day 1

SUMMARY:
Phase I study to evaluate the excretion of radioactivity, the metabolic profile, pharmacokinetics, safety and tolerability following a single oral administration of [14C] SPD557 in healthy male volunteers aged 18 to 50 years (inclusive).The purpose of this study is to investigate how and how quickly SPD557 or its break down products are excreted by analysing blood, faeces and urine samples collected during the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Males ages 18 to 50 years
* Have a body mass index (BMI) of ≥18.5 and ≤30 kg/m2
* Subject is willing to comply with any applicable contraceptive and sperm donation requirements

Key Exclusion criteria:

* Have participated in a [14C]-study within the last 6 months.
* Exposure to clinically significant radiation within 12 months prior to dose (for example, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring).
* Male subjects who consume more than 21 units of alcohol per week or 3 units per day.
* Subjects who report typically having more than 2 bowel movements per day, less than 3 bowel movements per week or those whose bowel habits have changed significantly within 30 days

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03-07 (Actual); Primary Completion 2013-04-12 (Actual); Study Completion 2013-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Covance, Madison, Wisconsin, United States

REFERENCES:
- [Result] Flach S, Croft M, Ding J, Budhram R, Pankratz T, Pennick M, Scarfe G, Troy S, Getsy J. Pharmacokinetics, absorption, and excretion of radiolabeled revexepride: a Phase I clinical trial using a microtracer and accelerator mass spectrometry-based approach. Drug Des Devel Ther. 2016 Sep 27;10:3125-3132. doi: 10.2147/DDDT.S107843. eCollection 2016. PMID 27729771

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiolabelled SSP-002358: A single oral dose of 2 mg radiolabeled SSP-002358 administered on Day 1
Period: Overall Study
Arm/Group | Radiolabelled SSP-002358
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiolabelled SSP-002358
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.5 (2.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 6

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC 0→∞) of Radiolabelled SSP-002358
Description: Area under the plasma concentration versus time curve from time 0 to infinity. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic (PK) Analysis Set included all subjects with at least 1 PK parameter estimated adequately in the Pharmacokinetic Concentration Analysis Set. Pharmacokinetic Concentration Analysis Set included all subjects who took at least 1 dose of investigational product and underwent plasma PK sampling and had evaluable PK assay results.
Measure: Mean (Standard Deviation); unit: pg*h/ml
Groups:
- Radiolabeled SSP-002358: A single oral dose of 2 mg radiolabeled SSP-002358 administered on Day 1
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
pg*h/ml | 43476 (13801)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Radiolabelled SSP-002358
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administered.
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
pg/ml | 4643 (894)

3. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
hours | 1.25 (1.17) [1.00 to 4.00]

4. Primary Outcome: Plasma Half-Life (T1/2) of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 5
hours | 11.0 (2.38)

5. Primary Outcome: AUC 0→∞ Whole Blood Total Radioactivity of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg equivalents*h/ml
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
pg equivalents*h/ml | 101960 (41581)

6. Primary Outcome: Cmax Whole Blood Total Radioactivity of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg equivalents/ml
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
pg equivalents/ml | 9252 (2138)

7. Primary Outcome: Tmax Whole Blood Total Radioactivity of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
hours | 2.00 [1.00 to 4.00]

8. Primary Outcome: Half-Life Whole Blood Total Radioactivity of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
hours | 6.96 (1.51)

9. Primary Outcome: AUC 0→∞ Plasma Total Radioactivity of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg equivalents*h/ml
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
pg equivalents*h/ml | 137314 (56101)

10. Primary Outcome: Cmax Plasma Total Radioactivity of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg equivalents/ml
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
pg equivalents/ml | 11658 (3538)

11. Primary Outcome: Tmax Plasma Total Radioactivity of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
hours | 1.50 [1.00 to 4.00]

12. Primary Outcome: Half-Life Plasma Total Radioactivity of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
hours | 10.9 (2.54)

13. Primary Outcome: Percent Total Radioactivity Excreted in Urine of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radioactivity
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
percentage of radioactivity | 38.2 (10.3)

14. Primary Outcome: Percent Total Radioactivity Excreted in Stool of Radiolabelled SSP-002358
Time Frame: Over 240 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radioactivity
Arm/Group | Radiolabeled SSP-002358
Number analyzed (Participants) | 6
percentage of radioactivity | 57.3 (10.4)

ADVERSE EVENTS:
Arm/Group | Radiolabelled SSP-002358
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiolabelled SSP-002358 (N=6)
Diarrhoea (Gastrointestinal disorders) | 5 (7)
Scratch (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.